CLINICAL TRIAL: NCT00076817
Title: A Phase I Double Blind Placebo Controlled Trial to Evaluate the Safety and Immunogenicity of the Aventis Pasteur ALVAC-HIV (vCP205) Administered to the Groin Area Versus the Deltoid Area
Brief Title: Safety and Effectiveness of Administering an HIV Vaccine in the Groin Versus the Arm
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 5R01AI050467-03 (NIH); UCLA MIG-003; 5R01AI050467-03 (NIH)
Record Dates: First submitted 2004-02-03; First posted 2004-02-06 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: HIV Preventive Vaccine; ALVAC Vaccine; Immunization Site; Deltoid; Groin; Targeted Inguinal Lymph Node; TILN
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Experimental): Participants will receive vaccine injections in the groin area or the upper arm
  Interventions: Biological: ALVAC-HIV (vCP205)
- 2 (Placebo Comparator): Participants will receive vaccine placebo injections in the groin area or the upper arm
  Interventions: Biological: ALVAC-HIV (vCP205)

INTERVENTIONS:
Biological: ALVAC-HIV (vCP205) — Canarypox virus vector vaccine
  Arms: 1
Biological: ALVAC-HIV (vCP205) — Canarypox virus vector vaccine placbo
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety of and immune system response to the ALVAC-HIV (vCP205) vaccine when it is injected either into the groin area or into the arm. The goal is to determine if injecting the vaccine into the groin area produces a better immune response in the lining of the rectum.

DETAILED DESCRIPTION:
HIV is most commonly transmitted via a mucosal surface. The mucosal lining is a potential site of both humoral and cellular protection through the activity of B lymphocytes, activated memory T lymphocytes, secretory IgA, and antigen presenting cells. In addition to systemic immunity, a preventive HIV vaccine should induce immune responses at the mucosal surfaces that are portals of HIV entry into the body.

Targeted lymph node immunization involves vaccine injection into the subcutaneous tissue near a lymph node. This strategy has proven effective in the simian immunodeficiency virus (SIV)/rhesus macaque model. The iliac and inguinal lymph nodes in the groin are the primary draining lymph nodes of the genitourinary and rectal tracts. This study will evaluate and compare the safety and immunogenicity of ALVAC-HIV (vCP205) when administered subcutaneously in the groin and intramuscularly in the deltoid region. ALVAC-HIV (vCP205) is a canarypox virus vector vaccine expressing portions of the gp120, Gag, and Pol genes.

Participants in this study will be randomly assigned to receive vaccine or placebo injections in the groin area or the upper arm. All participants will have three baseline visits for blood tests and sigmoidoscopies to measure baseline immune functions. After these visits, participants will receive weekly injections for 4 weeks. Groin injections will be given subcutaneously (under the skin) and upper arm injections will be given intramuscularly (into the muscle). Participants will have follow-up visits 5 and 11 months after the last immunization. Participants will have blood draws and sigmoidoscopies and will receive HIV risk reduction counseling throughout the study. Total length of participation will be approximately 14 months. Participants may continue to contact the study for HIV testing and study-related concerns for 1 year after study participation.

ELIGIBILITY:
Inclusion Criteria

* HIV uninfected
* Low risk for acquiring HIV-1 (no sexually transmitted disease within 1 year of study entry, no history of injection drug use, no sex with an HIV infected individual or active injection drug user within 6 months of study entry, no unsafe sexual activity with unknown partners) or mutually monogamous relationship with a known HIV seronegative partner (per report) for 6 months prior to study entry
* Willing to abstain from receptive anal intercourse during the 14 months of the study
* Available for follow-up during the 14 months of the study
* Acceptable methods of contraception

Exclusion Criteria

* Pregnant or lactating woman
* Allergy to eggs or neomycin
* Live attenuated vaccines within 60 days of study. Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) are not exclusionary, but should be given at least 1 month prior to study immunizations.
* Gastrointestinal complaints such as inflammatory bowel disease or chronic diarrhea
* Immunosuppression of any type, including those related to lupus, rheumatoid arthritis, leukemia, lymphoma, generalized malignancy, agammaglobulinemia, and therapy with alkylating agents, antimetabolites, or radiation
* Use of immunosuppressive medications within 6 months prior to study entry
* Thyroid disease
* Unstable asthma
* Exposure to or active tuberculosis
* Seizure disorders
* Bleeding disorders
* Splenectomy
* Hypertension (blood pressure less than 150/100 if on medication)
* Medical or psychiatric condition or occupational responsibilities which preclude participant's compliance with the study; specifically excluded are people with a history of suicide attempts, recent suicidal ideation, or who have past or present psychosis.
* Received HIV vaccines or placebo in a prior HIV vaccine trial
* Blood products within 120 days prior to study entry
* Immunoglobulin within 60 days prior to study entry
* Anaphylaxis or other serious adverse reactions to vaccines
* Serious allergic reaction to any substance requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension)
* Nonprescribed injection drug use
* Investigational research agents within 30 days prior to study entry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-06; Primary Completion 2007-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety of administering vCP205 vaccinations to healthy adult individuals | Throughout study

SECONDARY OUTCOMES:
Immunogenicity of SC vaccination with four doses of vCP205 administered in the groin area versus four doses administered IM in the deltoid region, as measured by CTL activity directed to canarypox and HIV-1 env, gag and pol gene products | Throughout study
Immunogenicity of SC vaccination with four doses of vCP205 administered in the groin area versus four doses administered IM in the deltoid region, as measured by anti-HIV-1 directed CD4+ T cell proliferative response to soluble p24 antigen | Throughout study
Immunogenicity of SC vaccination with four doses of vCP205 administered in the groin area versus four doses administered IM in the deltoid region, as measured by CD8+ T cell specificity for HIV-1 epitopes | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Anton, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for HIV and Digestive Diseases, Los Angeles, California, United States

REFERENCES:
- [Derived] Yang OO, Ibarrondo FJ, Price C, Hultin LE, Elliott J, Hultin PM, Shih R, Hausner MA, Ng HL, Hoffman J, Jamieson BD, Anton PA. Differential blood and mucosal immune responses against an HIV-1 vaccine administered via inguinal or deltoid injection. PLoS One. 2014 Feb 18;9(2):e88621. doi: 10.1371/journal.pone.0088621. eCollection 2014. PMID 24558403